CLINICAL TRIAL: NCT02320136
Title: Recording High Frequency Oscillations in Patients With Tumors and Epilepsy.
Acronym: HFO
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Other Study IDs: HFO
Record Dates: First submitted 2014-12-15; First posted 2014-12-19 (Estimated); Last update posted 2023-12-01 (Actual); Status verified 2023-11

CONDITIONS: Epilepsy; Tumor
MeSH Terms: conditions — Epilepsy; Neoplasms | interventions — Neuropsychological Tests

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- epilepsy: epilepsy patients
  Interventions: Behavioral: cognitive testing
- tumor with epilepsy: tumor patients with epileptic seizures
  Interventions: Behavioral: cognitive testing
- tumor without epilepsy: tumor patients without epileptic seizures
  Interventions: Behavioral: cognitive testing

INTERVENTIONS:
Behavioral: cognitive testing — patients perform simple tasks like watching a video or memorizing items

SUMMARY:
The investigators want to characterize high-frequency oscillations (HFOs) in intracranial recordings, which may occur as markers of epileptogenic tissue and also under physiological stimulation.

The investigators want to show that recording of high-frequency oscillations (HFOs) is feasible in our project population both intraoperatively and during presurgical physiological conditions.

ELIGIBILITY:
Inclusion Criteria:

* Patients intend to be treated at the Klinik für Neurochirurgie
* Patients fall into one of the patient groups: (1) Patients with symptomatic epilepsy with focal and/or secondary generalized seizures resistant to medication where a neurosurgical resection is considered as an intervention of epilepsy surgery. (2)Patients where a tumor is planned to be resected that has caused preoperative seizures. (3) Patients where a tumor is planned to be resected that has not caused preoperative seizures.
* Male and Female subjects 18 years to 99 years of age
* Written informed consent after participants' information

Exclusion Criteria:

* contraindications on ethical grounds
* known or suspected non-compliance, drug or alcohol abuse,
* enrolment into a clinical trial within last 4 weeks

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 1. Patients with epilepsy where a surgical resection is considered.
  2. Patients where a tumor will be resected that has caused preoperative seizures.
  3. Patients where a tumor will be resected that has not caused preoperative seizures.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2014-06; Primary Completion 2024-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
HFO (high-frequency oscillations) occurrence | 1 week

CONTACTS AND LOCATIONS:
Overall Officials: Johannes Sarnthein, Prof Dr, Principal Investigator — Universitätsspital Zürich